CLINICAL TRIAL: NCT00457756
Title: The Effect of an Integrative Dietary Supplement on the Lipid Profile of Subjects With Hypercholesterolemia
Brief Title: The Effect of BiosLife on Serum Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Unicity International (Unknown)
Responsible Party: Paul Hopkins, MD, MSPH, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BiosLife 2005-4
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2008-05

CONDITIONS: Hypercholesterolemia
Keywords: LDL cholesterol; HDL cholesterol; natural supplement; guar gum; phytosterols; policosanol; chrysanthemum
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Active Comparator): Cohort I subjects will take supplement for 12 weeks
  Interventions: Dietary Supplement: BiosLife Complete
- II (Placebo Comparator): Cohort II will take placebo for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: BiosLife Complete
  Arms: I
Dietary Supplement: Placebo
  Arms: II

SUMMARY:
This is a double-blind, placebo-controlled study to assess the effectiveness of BiosLife in lowering serum LDL cholesterol and raising HDL cholesterol. BiosLife is a natural supplement (mixed in water and taken twice daily) which contains guar gum and other natural soluble fibers, phytosterols, policosanol, and a proprietary chrysanthemum extract. Approximately 100 subjects with baseline LDL cholesterol of 110-190 mg/dL will be randomized in a 2:1 ratio to BiosLife or a look-alike placebo. Changes in lipids from baseline will be assessed at 6 weeks and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* LDL-C 110 - 190 mg/dL
* For current lipid-lowering prescription therapy users, the dose of lipid-lowering medication must have been constant for 3 months with no current plan for change in dose.
* Age 18 - 85 years

Exclusion Criteria:

* Type 1 diabetes
* Severe hypertension, defined as at least 180 / 100 mmHg
* Any other health condition that may interfere with the study results, as judged by the principle investigator
* Allergy against any of the ingredients in the tested product
* Any medical condition, in which fiber consumption is contraindicated (e.g. Crohn's disease
* The use of nutritional supplements during the last two months containing one or more similar ingredients, as the tested supplement.
* History of alcohol or drug abuse, psychological or other mental issues that are likely to invalidate informed consent, or limit the ability of the patient to comply with the protocol requirements
* Participation in any other studies involving investigational or marketed product concomitantly or within one month prior to entry into the study
* Pregnant or breast feeding
* Persons who eat only 1 meal per day

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol | 12 weeks
HDL cholesterol | 12 weeks

SECONDARY OUTCOMES:
triglycerides | 12 weeks
LDL particle number | 12 weeks
LDL particle size distribution | 12 weeks
HDL particle number | 12 weeks
HDL particle size distribution | 12 weeks
VLDL particle number | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul N Hopkins, MD, MSPH, Principal Investigator — University of Utah
Locations (1):
- Cardiovascular Genetics, University of Utah, 420 Chipeta Way, Room 1160, Salt Lake City, Utah, United States